CLINICAL TRIAL: NCT05649618
Title: A Single-center, Open-label Clinical Study of TIL Cells for the Treatment of the Recurrent/Metastatic Solid Tumors Patients Who Had Failed Standard Therapy
Brief Title: TIL Cells for the Treatment of the Advanced Solid Tumors Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJ001
Record Dates: First submitted 2022-10-26; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Solid Tumor
MeSH Terms: interventions — fludarabine; Cyclophosphamide; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor Infiltrating Lymphocytes (Experimental): TIL cells (2.5×10^9-5×10^10) will be infused i.v. to patients with advanced solid tumors after non-myeloablative lymphocyte-depleting preparative regimen.
  Interventions: Biological: Tumor Infiltrating Lymphocytes; Drug: Fludarabine; Drug: Cyclophosphamide Capsules; Drug: IL-2

INTERVENTIONS:
Biological: Tumor Infiltrating Lymphocytes — On day 0 patients will be intravenous infusion of TILs
Drug: Fludarabine — Part of the non-myeloablative lymphocyte-depleting preparative regimen
Drug: Cyclophosphamide Capsules — Part of the non-myeloablative lymphocyte-depleting preparative regimen.
Drug: IL-2 — Following cell infusion, the patient receives high-dose bolus IL-2, which is dosed to individual patient tolerance.

SUMMARY:
This study is to investigate the safety and efficacy of tumor infiltrating lymphocyte (TILs) therapy in patients with Advanced malignant solid tumors. TILs are expanded from tumor resections or biopsies, and after ex vivo stimulation, activation and extensive expansion, are reinfused to patients after non-myeloablative lymphocyte-depleting preparative regimen.

DETAILED DESCRIPTION:
This is a single-center, open-label, Phase I clinical study of TILs for the treatment of the recurrent/metastatic solid tumors patients who had failed standard therapy.

TILs are expanded from tumor resections or biopsies, and after ex vivo stimulation, activation and extensive expansion, are reinfused to patients after non-myeloablative lymphocyte-depleting preparative regimen.

The primary purpose of this study is to evaluate the safety and tolerability of TILs in patients with recurrent/metastatic solid tumors.

The second purpose of this study is to preliminarily explore the effectiveness of TILs in patients with recurrent/metastatic solid tumors.

Eligibility:

Adults aging 18-75 who were failed to standard treatment or have no standard treatment with recurrent/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Have the willingness to communicate with investigator, be able to understand and follow the trail requirements, and voluntarily to participate in the trail;
2. 18 ~ 75 years;
3. The expected survival period is at least 3 months;
4. ECOG score of 0-1;
5. There is at least one lesion that can be operated or biopsied for the preparation of TIL;
6. According to RECIST 1.1 standard, there is at least one measurable target lesion for efficacy evaluation;
7. Patients with recurrent or metastatic solid tumors confirmed by histopathology;
8. Subjects who failed standard treatment in the past or have no standard treatment currently tor who are judged by the investigator to be unsuitable for current standard treatment for other reasons, and the objective imaging assessment is disease progression

Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding, or have a positive blood pregnancy test at baseline ;
2. Subjects who have had severe allergic reactions to any drug or its components in this trial in the past;
3. Subjects who have received any investigational drug within 28 days before the infusion of TIL cells, or participated in another clinical study at the same time;
4. Subjects who have other known history of malignant tumors in the past 5 years, except for localized tumors that have been cured, including in situ cervical carcinoma, basal cell carcinoma of the skin, and in situ prostate carcinoma;
5. Patients who have received adoptive cell therapy in the past;
6. According to the judgment of the investigator, the condition of the subject is not suitable for this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-12-05 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | up to Day 28
  Dose Limiting Toxicity (DLT) is defined as patients with the adverse event (AE) or laboratory abnormality recognized by Investigators, and should be possibly related to TILs therapy.
Adverse Event | up to 24 months
  The severity and incidence of various adverse events and serious adverse events

SECONDARY OUTCOMES:
Overall response rate(ORR) | up to 24 months
Progression free survival (PFS) | up to 24 months
Overall survival (OS) | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: zhiyong He, Principal Investigator — Fujian Cancer Hospital

IPD SHARING:
Plan to Share IPD: No